CLINICAL TRIAL: NCT05212168
Title: A Phase 2b Double-Blinded, Randomized, Placebo-Controlled, Human Norovirus GI.1 (Norwalk Virus Inoculum) Challenge Study Following Administration of an Oral, Single-dose Norovirus Vaccine Expressing GI.1 VP1 and dsRNA Adjuvant to Protect Against Norovirus Gastroenteritis (NVG) in Healthy Adult Volunteers
Brief Title: Norovirus Challenge Study
Acronym: G1-1 Challenge
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: VXA-NVV-201
Record Dates: First submitted 2022-01-25; First posted 2022-01-27 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-09

CONDITIONS: Norovirus Infections
MeSH Terms: conditions — Caliciviridae Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Vaccine Arm (Active Comparator): Subjects receiving Norovirus GI.1 Norwalk VP1 Vaccine, Oral E1-/E3-Deleted Replication Defective Recombinant Adenovirus 5 with dsRNA Adjuvant
  Interventions: Biological: VXA-G1.1-NN; Biological: Norovirus GI.1 Norwalk Virus Inoculum
- Placebo Arm (Placebo Comparator): Subject receiving Placebo oral tablets similar in appearance and number to active vaccine tablets
  Interventions: Other: Placebo Tablets; Biological: Norovirus GI.1 Norwalk Virus Inoculum

INTERVENTIONS:
Biological: VXA-G1.1-NN — Norovirus GI.1 Norwalk VP1 Vaccine, Oral E1-/E3-Deleted Replication Defective Recombinant Adenovirus 5 with dsRNA Adjuvant
  Arms: Active Vaccine Arm
Other: Placebo Tablets — Oral tablets similar in appearance and number to active vaccine tablets
  Arms: Placebo Arm
Biological: Norovirus GI.1 Norwalk Virus Inoculum — Norwalk Virus Inoculum Lot 01-09NV

SUMMARY:
This is a Phase 2b randomized, double-blind, placebo-controlled vaccination and challenge study to assess the protective efficacy of the Vaxart Norovirus vaccine (VXA-G1.1-NN). Healthy adults will be randomized in a 1:1 ratio to receive one oral dose of vaccine or placebo.

* Arm 1: VXA-G1.1-NN oral vaccine tablets [1x1011 IU±0.5 log]
* Arm 2: Placebo tablets similar in appearance and number to active vaccine tablets

Approximately 28 days post-vaccination, subjects will be admitted to an isolation ward and challenged with the NV GI.1 Norwalk challenge strain. After challenge, subjects will be monitored for signs and symptoms of acute gastroenteritis (AGE) from Day 29 to discharge. At 4 days post challenge (Day 33) asymptomatic subjects will be discharged from the isolation ward and will be followed in a series of outpatient visits and telephone calls. Symptomatic subjects may be kept in the isolation ward for up to an additional 3 days.

DETAILED DESCRIPTION:
Study Population Healthy male and female adult volunteers age 18 to 49 years inclusive with blood type O or A and who are confirmed H type-1 antigen secretory positive Investigational Product

Active Vaccine:

* Norovirus GI.1 Norwalk VP1 Vaccine (VXA-G1.1-NN), an Oral E1/E3-Deleted Replication-Defective Recombinant Adenovirus serotype 5 with double-stranded ribonucleic acid (dsRNA) Adjuvant. The vaccine vector encodes for a full-length VP1 gene from Norwalk virus (NV). The adjuvant is a short hairpin RNA, expressed as a 21 nucleotide sequence (GAAACGA TATGGGCTGAATAC) as a tandem sequence in forward and reverse orientations separated by 6 nucleotides that comprise the loop of the RNA. The final drug product (DP) is formulated into enteric-coated tablet.
* Dose: 1x10E11 IU±0.5 log

Placebo Control:

• Oral tablets similar in appearance and number to active vaccine tablets Multiple tablets of study drug will be dispensed to allow delivery of the intended vaccine dose (1x10E11 IU). A matching number of placebo tablets will be dispensed to maintain the study blinding.

Viral Challenge Inoculum

* Norovirus GI.1 (Norwalk Virus Inoculum Lot 001-09NV, IND 14697)
* Dose: 1x10E6 Genomic Copies (GC). A dose which allows 50% - 65% infectivity in the healthy adult population (per NV infection rate observed in the GI.1 viral titration study

Study Hypothesis Norovirus vaccine (VXA-G1.1-NN) will protect against Norovirus Gastroenteritis (NVG) related to norovirus (NoV) infection in the challenge model

Approximately 120 subjects will be dosed in the vaccination phase to ensure at least 100 subjects (~ 50 VXA-G1.1-NN vaccine and 50 placebo) are available to participate in the challenge phase. Approximately 28 days post-vaccination, subjects will be admitted to an isolation ward and challenged with the NV GI.1 Norwalk challenge strain. After challenge, subjects will be monitored for signs and symptoms of acute gastroenteritis (AGE) from Day 29 to discharge. NV illness lasts 2-4 days and is self-limited. At 4 days post challenge (Day 33) asymptomatic subjects will be discharged from the isolation ward and will be followed in a series of outpatient visits and telephone calls. Symptomatic subjects may be kept in the isolation ward for up to an additional 3 days.

The following study visits and remote contacts will be conducted during the study

Vaccination Phase:

* Pre-Screening Period (Days -90 to Screening) may be utilized for purposes of ascertaining subjects' H type-1 antigen secretory status and blood type
* Screening Period (Days -45 to -1)
* Day 1 Visit (Baseline assessments; day of randomization and vaccination)
* Day 8 Visit (safety and evaluation of immune response)
* Day 28 (evaluation of immune response; 1 day prior to challenge, start inpatient stay)

Challenge Phase:

* Day 29 (viral challenge, sequestration)
* Days 30 to 33 (sequestration - discharge; +3 days)
* Day 36 Visit (evaluation of immune response and safety assessment)
* Day 57 Visit (end of active period)

Safety Follow-Up:

* Day 120, Day 180, Day 240 and Day 300 (follow-up contact)
* Day 185 (follow-up phone call): Study completion

An independent Safety Monitoring Committee (SMC) will convene at pre-defined intervals during the norovirus challenge period, and also ad hoc as needed during the vaccination and challenge periods, to oversee the safety of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 - 49 years, inclusive
2. Able to give written informed consent
3. Healthy, as determined by the principal investigator (PI) or PI in consultation with the research monitor and Sponsor Healthy = No clinically significant health concerns or medical illness, as determined by medical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratories (complete blood count (CBC), chemistry and urinalysis)
4. Comprehension of the study requirements with ability and willingness to complete all assessments and comply with confinement period post viral challenge, and all scheduled visits and contacts
5. Confirmed blood type (A or O)
6. Demonstrated to be H type-1 antigen secretor positive (by saliva test)
7. Body mass index between 17 and 35 kg/m2, inclusive, at Screening
8. Female participants must have a negative pregnancy test at pre-vaccination and pre-challenge and fulfill one of the following Criteria:

   1. At least one year post-menopausal;
   2. Surgically sterile;
   3. Use of oral, implantable, transdermal or injectable contraceptives for 30 days prior to immunization and until 60 days after challenge;

   i. A reliable form of contraception must be approved by the Investigator (eg, double barrier method, Depo-Provera, intrauterine device, Norplant, oral contraceptives, contraceptive patches) d. Not be sexually active (abstinent) or in a same sex relationship (must be discussed with site staff and documented)
9. Male subjects must agree not to father a child or donate sperm, as well as to use contraception/barrier (a male condom) or be abstinent from heterosexual intercourse, from vaccination through the active period (Day 57)

Exclusion Criteria:

1. Administration/use of any investigational drug or device 30 days prior to vaccination through the active period (Day 57)
2. Administration of any licensed vaccine within 30 days prior to vaccination or planned use of the above stated during the active period (through Day 57)
3. Presence of a significant medical condition, which, in the opinion of the investigator, precludes participation in the study. Significant medical condition = for example, psychiatric conditions, or gastrointestinal disease, such as peptic ulcer, symptoms or evidence of active gastritis or gastroesophageal reflux disease, inflammatory bowel disease, alcohol or illicit drug abuse/dependency, or other laboratory abnormalities
4. Laboratory values outside the range of normal for platelet counts and the following coagulation tests: prothromibin time test (PT/INR), activated partial thromboplastine time test (aPTT) and fibrinogen
5. Any of the following history or conditions that may lead to higher risk of clotting events and/or thrombocytopenia:

   1. Family or personal history of bleeding or thrombosis
   2. History of heparin-related thrombotic events, and/or receiving heparin treatments
   3. History of autoimmune or inflammatory disease
   4. Presence of any of the following conditions known to increase risk of thrombosis within 6 months prior to screening:

      * Recent surgery other than removal/biopsy of cutaneous lesions
      * Immobility (confined to bed or wheelchair for 3 or more successive days)
      * Head trauma with loss of consciousness or documented brain injury
      * Receipt of anticoagulants for prophylaxis of thrombosis
      * Recent clinically significant infection
6. Any one of the following ECG findings within 45 days prior to vaccination:

   Exclusionary ECG findings:
   1. QTc F (interval duration > 450 msec (male) or > 470 msec (female)
   2. QRS interval greater than 120 msec
   3. PR interval greater than 220 msec
   4. Clinically significant ST-T wave changes or pathologic Q waves
7. History of cancer or cancer treatment within past 3 years (excluding basal cell or squamous cell carcinomas)
8. Presence of immunosuppression or medical condition possibly associated with impaired immune responsiveness, including diabetes mellitus or angioedema
9. Donation or use of blood or blood products within 30 days prior to vaccination through the active period (Day 57)
10. Diagnosed bleeding disorder or significant bruising or bleeding difficulties that could make blood draws problematic
11. Any condition that resulted in the absence or removal of the spleen
12. Evidence of confirmed infection with human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) with confirmatory assays
13. Abnormal stool pattern (fewer than 3 bowel movements per week or more than 3 per day)
14. History of irritable bowel disease or inflammatory digestive or gastrointestinal condition that could affect the distribution / safety evaluation of an orally administered vaccine targeting the mucosa of the small intestine.

    Such conditions may include but are not limited to:
    1. Esophageal Motility Disorder
    2. Malignancy
    3. Malabsorption (e.g. Celiac disease, gluten intolerance)
    4. Pancreaticobiliary disorders
    5. Irritable bowel syndrome
    6. Inflammatory Bowel Disease
    7. Surgical Resection with the exception of appendectomy or a minor resection that is deemed acceptable by investigator and sponsor
    8. Gastroesophageal reflux disease (GERD)
    9. Hiatal Hernia
    10. Peptic Ulcer (History of cholecystectomy is not exclusionary)
15. Use of proton pump inhibitors, H2 blockers or antacids within 7 days prior to vaccination through the active period (Day 57)
16. Use of antibiotics within 30 days prior to vaccination through the active period (Day 57) Note: use of a brief (≤ 10 days) course of oral or topical antibiotic for minor upper respiratory infection (URI), urinary tract infection (UTI), dental work, or skin infection allowed within the screening period, but must be completed 7 days prior to first vaccination
17. Use of medication known to affect the immune function (e.g. systemic corticosteroids and others) within 14 days prior to vaccination through the active period (Day 57)
18. Regular use of nonsteroidal anti-inflammatory drugs within 7 days prior to vaccination through the active period (Day 57)
19. Use of over-the-counter probiotics or antidiarrheals within 7 days prior to vaccination through the active period (Day 57)
20. Evidence of recent (within 2 months of vaccination) or of current nonbacterial gastroenteritis suggestive of NV infection [vomiting or unformed or watery stools (> 2 during a 24-hour period)]
21. Any gastroenteritis within the past 2 weeks prior to vaccination
22. Acute disease within 72 hours prior to vaccination, defined as the presence of a moderate or severe illness with or without fever (as determined by the Investigator through medical history and physical examination). (Assessment may be repeated during screening period)
23. Presence of a fever ≥ 38ºC measured orally at baseline
24. History if hematochezia (blood in stool) or melena (black stool)
25. Any significant hospitalization within the last year which in the opinion of the investigator or sponsor could interfere with study participation
26. History of serious reactions to any vaccination such as anaphylaxis, respiratory problems, Guillain-Barre syndrome, hives or abdominal pain
27. History of a hypersensitivity or allergic reaction to any component of the investigational vaccine or placebo, including but not limited to fish gelatin. Subjects with known fish allergies should be excluded.
28. History of drug, alcohol or chemical abuse within 1 year prior to vaccination
29. Positive test for drugs of abuse or alcohol at screening, vaccination baseline and pre-challenge (except for previous marijuana use; concurrent or ongoing use of marijuana during the active study period).
30. Consistent/habitual smoking within 2 months prior to vaccination (defined as smoking ≥ 1 pack of cigarettes a day). Smoking is not permitted during the inpatient stay
31. Other conditions, in the clinical judgment of the investigator, that would jeopardize the safety or rights of a subject or interfere with the evaluation of the study

    Social/Occupational:
32. Living with or having daily contact with children < 5 years old or women known to be pregnant or nursing; this includes significant contact at home, school, day-care, or equivalent facilities
33. Living with or having daily contact with elderly persons > 70 years of age or infirmed, diapered individuals, persons with disabilities or incontinence; this includes at work or visits to nursing homes and day-care or equivalent facilities
34. Employment in the food service industry such as restaurant or cafeteria facilities; specifically, this includes persons whose employment requires food handling and processing in the 4 weeks following viral challenge
35. Health-care workers with patient contact expected in the 4 weeks following viral challenge
36. Expected contact, via employment or at home, with immunocompromised persons in the 4 weeks following viral challenge. Immunocompromised persons = HIV-positive, receiving immunosuppressive medications such as oral steroids, anti-neoplastic agents
37. Presence of household members who have received the Ad4 or Ad7 vaccines within 2 months prior to vaccination
38. Employment as an airline flight attendant or cruise ship crew, scheduled to work in the 4 weeks following challenge
39. Persons planning to live in a confined environment (eg, a cruise, camp, etc.) in the 4 weeks following viral challenge

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Cummings, MD, Study Director — Vaxart, Inc.
Locations (1):
- AltaSciences LA, Cypress, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 center in the United States (US) between December 2021 and October 2023.
Pre-assignment Details: Healthy participants were randomized in a 1:1 ratio to receive a single oral dose of VXA-G1.1-NN or placebo. The total study duration for each participant was approximately 16 months, including screening, a 28-day vaccination phase, a 28-day Challenge Phase, and up to 365 days of safety follow-up.
Groups:
- VXA-G1.1-NN: Healthy participants received a single dose of VXA-G1.1-NN oral vaccine tablet. Approximately 29 days post-vaccination, participants began the Challenge Phase Day 1. During this phase, participants were isolated, exposed to the Norwalk virus (NV) genogroup I genotype 1 (GI.1) Norwalk challenge strain, and monitored for signs and symptoms of acute gastroenteritis (AGE) until discharge. Asymptomatic participants were discharged on Day 3 of the Challenge Phase and continued with a series of outpatient visits and telephone follow-ups. Symptomatic participants could remain in isolation for up to an additional 3 days.
- Placebo: Healthy participants received a single dose of matching placebo. Approximately 29 days post-vaccination, participants began the Challenge Phase Day 1. During this phase, participants were isolated, exposed to the NV GI.1 Norwalk challenge strain, and monitored for signs and symptoms of AGE until discharge. Asymptomatic participants were discharged on Day 3 of the Challenge Phase and continued with a series of outpatient visits and telephone follow-ups. Symptomatic participants could remain in isolation for up to an additional 3 days.
Period: Overall Study
Arm/Group | VXA-G1.1-NN | Placebo
Started (Participants who received interventions during the vaccination phase.) | 86 | 79
Entered Challenge Phase | 76 | 65
Completed | 52 | 42
Not Completed | 34 | 37
Not completed — Lost to Follow-up | 0 | 3
Not completed — Study terminated by sponsor | 30 | 27
Not completed — Other | 4 | 7

BASELINE CHARACTERISTICS:
Population: Full Analysis Population (FAP): all randomized participants analyzed by randomized vaccination group assignment, who received study vaccination (active or placebo), and had available data for the specified analysis.
Groups:
- VXA-G1.1-NN: Healthy participants received a single dose of VXA-G1.1-NN oral vaccine tablet. Approximately 29 days post-vaccination, participants began the Challenge Phase Day 1. During this phase, participants were isolated, exposed to the NV GI.1 Norwalk challenge strain, and monitored for signs and symptoms of AGE until discharge. Asymptomatic participants were discharged on Day 3 of the Challenge Phase and continued with a series of outpatient visits and telephone follow-ups. Symptomatic participants could remain in isolation for up to an additional 3 days.
- Total: Total of all reporting groups
Arm/Group | VXA-G1.1-NN | Placebo | Total
Number analyzed (Participants) | 86 | 79 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (8) | 34 (7) | 35 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 31 | 74
  Male | 43 | 48 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 33 | 70
  Not Hispanic or Latino | 49 | 46 | 95
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 8 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 14 | 35
  White | 54 | 54 | 108
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Norovirus Gastroenteritis (NVG)
Description: NVG is a composite endpoint defined as meeting both the definition of AGE and NV.
  AGE was defined as meeting any one of 3 criteria (diarrhea, vomiting, or diarrhea and vomiting) in any 24-hr rolling period. The individual criteria for diarrhea, vomiting, or diarrhea and vomiting were as follows:
  1. Diarrhea: i. ≥ 3 loose or liquid stools in any 24-hr rolling period, or ii. 400 g of loose or liquid stools in any 24-hr rolling period 2. Vomiting: ≥ 2 vomiting episodes in any 24-hr rolling period, or 3. Diarrhea and vomiting: i. one vomiting episode plus any loose or liquid stool in any 24-hr rolling period ii. one vomiting episode plus ≥ 2 of the following events in any 24-hr rolling period:
  1. nausea
  2. fever (oral temperature ≥ 37.6°C)
  3. abdominal cramps or pains
  4. abdominal gurgling or bloating
  5. myalgia NV infection was defined as having 1 or more positive results in stool or urine by quantitative real time reverse transcription polymerase chain reaction (qRT-PCR).
Time Frame: Up to approximately Day 57
Population: FAP: all randomized participants analyzed by randomized vaccination group assignment, who received study vaccination (active or placebo), and had available data for the specified analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 76 | 65
Participants | 34 | 37

2. Primary Outcome: Levels of Viral Protein 1, Major Capsid, or Surface Protein of Viruses (VP1)-Specific Immunoglobulin A (IgA) Antibody-Secreting Cell (ASC) Against Norwalk at Day 8
Description: Blood samples were collected at different timepoints throughout the study.
Time Frame: Day 8
Population: Immunogenicity Population: all randomized participants who received study vaccination (active or placebo), and had available data for the specified analysis.
Measure: Mean (95% Confidence Interval); unit: cells/10^6 PBMCs
Groups:
- VXA-G1.1-NN: Healthy participants received a single dose of VXA-G1.1-NN oral vaccine tablet. Approximately 29 days post-vaccination, participants began the Challenge Phase Day 1. During this phase, participants were isolated, exposed to the NV GI.1 Norwalk challenge strain, and monitored for signs and symptoms of AGE until discharge. Asymptomatic participants were discharged on Day 3 of the Challenge Phase and continued with a series of outpatient visits and telephone follow-ups. Symptomatic participants could remain in isolation for up to an additional 3 days. The total duration of participation in the study for each participant was approximately 16 months and included a safety follow-up for up to 365 days.
- Placebo: Healthy participants received a single dose of matching placebo. Approximately 29 days post-vaccination, participants began the Challenge Phase Day 1. During this phase, participants were isolated, exposed to the NV GI.1 Norwalk challenge strain, and monitored for signs and symptoms of AGE until discharge. Asymptomatic participants were discharged on Day 3 of the Challenge Phase and continued with a series of outpatient visits and telephone follow-ups. Symptomatic participants could remain in isolation for up to an additional 3 days. The total duration of participation in the study for each participant was approximately 16 months and included a safety follow-up for up to 365 days.
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 83 | 79
cells/10^6 PBMCs | 79.5 [69.2 to 87.6] | 0 [0.0 to 4.6]

3. Primary Outcome: Geometric Mean Titer (GMT) of Histo-blood Group Antigen (HBGA) Blocking Antibodies Against NV by Blocking Titer 50 (BT50) at Day 28
Description: Blood samples were collected at different timepoints throughout the study. A positive change indicates an increase in titers.
Time Frame: Day 28
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 82 | 71
Geometric mean titer | 131.6 [101.2 to 171.2] | 33.2 [26.4 to 41.8]

4. Primary Outcome: VP1-specific Serum Immunoglobulin G (IgG) Response at Day 28
Description: Blood samples were collected at different timepoints throughout the study.
Time Frame: Day 28
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 82 | 71
AU/mL | 4413573.1 [3167431.7 to 6149975.6] | 700657.0 [508361.8 to 965690.5]

5. Primary Outcome: VP1-specific Serum IgA at Day 28
Description: Blood samples were collected at different timepoints throughout the study.
Time Frame: Day 28
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 82 | 71
AU/mL | 5555338.7 [3713874.2 to 8309863.5] | 670496.0 [450873.7 to 997097.1]

6. Secondary Outcome: Number of Participants Who Experienced Solicited Symptoms of Reactogenicity
Description: Solicited symptoms of reactogenicity included:
  * Gastrointestinal reactions: nausea, vomiting, diarrhea and abdominal pain
  * Systemic reactogenicity: malaise/fatigue, anorexia, fever, headache and myalgia
Time Frame: Up to Day 8
Population: Safety Population: consisted of all participants who received any study vaccination (active or placebo). This population was summarized according to the actual vaccination received.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 86 | 79
Participants | 50 | 36

7. Secondary Outcome: Number of Participants Who Experienced Unsolicited Adverse Events (AEs) During the Vaccination Phase
Description: Unsolicited AEs referred to any AEs that occurred during a clinical trial but were not specifically pre-defined or actively sought by the study protocol. Unsolicited AEs could include any medical condition or symptom, whether or not it was related to the intervention being studied.
Time Frame: Up to Day 28 of Vaccination Phase (28-days phase)
Population: Vaccination Phase Safety Population: consisted of all participants who received any study vaccination (active or placebo). This population was summarized according to the actual vaccination received.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 86 | 79
Participants | 7 | 9

8. Secondary Outcome: Number of Participants Who Experienced Serious AEs (SAEs), AEs of Specific Interest (AESIs), and New Onsets of Chronic Illness (NOCIs)
Description: A SAE was any AE that resulted in one or more of the following outcomes: death, a life-threatening event where the subject was at immediate risk of death (not hypothetically), inpatient hospitalization or the prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of normal life functions, congenital abnormality or birth defect, or an important medical event that, that jeopardized the participant's health or required medical or surgical intervention to prevent a serious outcome. A NOCI was defined as the diagnosis post-study drug administration of a new medical condition, which was chronic in nature, including those potentially controllable by medication (e.g., diabetes, asthma).
Time Frame: Up to approximately 12 months post vaccination
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 86 | 79
Participants
  All SAEs | 0 | 1
  All AESI | 0 | 1
  All NOCI | 0 | 0

9. Secondary Outcome: Number of Participants Who Experienced Unsolicited AEs During the Challenge Phase
Description: as for outcome 7
Time Frame: Up to Day 29 of Challenge Phase (28-days phase)
Population: Challenge Phase Safety Population: consisted of all participants who received any study vaccination (active or placebo) and entered the 28-days Challenge Phase. This population was summarized according to the actual vaccination received.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 76 | 65
Participants | 31 | 23

10. Secondary Outcome: Number of Participants With AGE During the Inpatient Challenge Phase
Description: AGE was defined as meeting any one of 3 criteria (diarrhea, vomiting, or diarrhea and vomiting) in any 24-hr rolling period. The individual criteria for diarrhea, vomiting, or diarrhea and vomiting were as follows:
  1. Diarrhea: i. ≥ 3 loose or liquid stools produced in any 24-hr rolling period, or ii. 400 g of loose or liquid stools produced in any 24-hr rolling period 2. Vomiting: ≥ 2 vomiting episodes in any 24-hr rolling period, or 3. Diarrhea and vomiting: i. one vomiting episode plus any loose or liquid stool in any 24-hr rolling period ii. one vomiting episode plus ≥ 2 of the following events in any 24-hr rolling period:
  1. nausea
  2. fever (oral temperature ≥ 37.6°C)
  3. abdominal cramps or pains
  4. abdominal gurgling or bloating
  5. myalgia
Time Frame: Day 28 of Challenge Phase (28-days phase)
Population: Challenge Phase FAP: consisted of all participants who received any study vaccination (active or placebo) and entered the 28-days Challenge Phase. This population was summarized according to the actual vaccination received.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 76 | 65
Participants | 40 | 39

11. Secondary Outcome: Severity of AGE Assessed Using the Modified Vesikari Scale
Description: The Modified Vesikari Scale is a tool used to assess the severity of AGE by evaluating symptoms such as diarrhea, vomiting, fever, and dehydration. It scores these symptoms based on their frequency and severity, with a minimum score of 0 and a maximum score of 20, where higher scores indicate more severe symptoms and lower scores suggest milder or no symptoms and severity.
Time Frame: Up to approximately Day 36
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 76 | 65
Score on scale | 4.2 [3.5 to 4.8] | 4.4 [3.8 to 5.1]

12. Secondary Outcome: Number of Participants Who Experienced Moderate or Severe Gastroenteritis
Description: Moderate or severe gastroenteritis was defined by cumulative loose stools ≥ 1000gr during the inpatient period.
Time Frame: Up to approximately Day 57
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 76 | 65
Participants | 14 | 7

13. Secondary Outcome: Duration of AGE
Description: Time to onset of AGE was calculated as the time from challenge administration to the first recorded instance of an event satisfying the criteria for AGE.
  AGE was defined as meeting any of the 3 criteria:
  1. Diarrhea: i. ≥ 3 loose or liquid stools in any 24-hr rolling period, or ii. 400 g of loose or liquid stools in any 24-hr rolling period 2. Vomiting: ≥ 2 vomiting episodes in any 24-hr rolling period, or 3. Diarrhea and vomiting: i. one vomiting episode plus any loose or liquid stool in any 24-hr rolling period ii. one vomiting episode plus ≥ 2 of the following events in any 24-hr rolling period:
  1. nausea
  2. fever (oral temperature ≥ 37.6°C)
  3. abdominal cramps or pains
  4. abdominal gurgling or bloating
  5. myalgia
Time Frame: Up to approximately Day 57
Population: Challenge Phase FAP: consisted of all participants who received any study vaccination (active or placebo) and entered the 28-days Challenge Phase. This population was summarized according to the actual vaccination received. Only AGE positive participants were included in the analysis
Measure: Median (Full Range); unit: Hours
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 76 | 65
Hours | 59.0 [26.7 to 117.3] | 55.8 [28.6 to 107.1]

14. Secondary Outcome: Number of Participants Who Experienced Incidences of Diarrhea or Emesis
Description: Classification of diarrhea was done through grading stools with Grade 3 (thick liquid stool) to Grade 5 (clear water diarrheal stool) being considered diarrhea.
Time Frame: Up to approximately Day 57
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 76 | 65
Participants
  Diarrhea | 52 | 44
  Emesis | 28 | 33

15. Secondary Outcome: Number of Participants With Norovirus (NoV) Infection up to Challenge Period Day 8
Description: NoV infection was defined as a positive qRT-PCR in stool or emesis up to Challenge Period Day 8, and the presence of NV antigen in stool.
Time Frame: Challenge Phase Day 8 (equal to Study Day 36)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 76 | 65
Participants | 44 | 53

16. Secondary Outcome: Geometric Mean Genome Copies (GCs) of NoV Shedding in Stool Measured by qRT-PCR
Description: NoV shedding was assessed by qRT-PCR. Stool samples were reported on 10^3 copies/gm. If a participant produced multiple results for a given study day, the result with the largest shedding response was used for analysis. Samples that were reported as "Not Quantifiable" or as lower than the limit of detection (LOD) were analyzed as ½2*LOD (76.2).
Time Frame: Pre-challenge up to Day 8 of Challenge Phase (equal to Study Day 36)
Population: Challenge Phase FAP: consisted of all participants who received any study vaccination (active or placebo) and entered the 28-days Challenge Phase. This population was summarized according to the actual vaccination received. Only participants with available data at each time point were included.
Measure: Geometric Mean (95% Confidence Interval); unit: 10^3 copies/gm
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 82 | 72
10^3 copies/gm
  Pre-challenge | 76.2 [NA to NA] — The 95% confidence interval was not estimable as all samples were below the LOD. | 76.2 [NA to NA] — The 95% confidence interval was not estimable as all samples were below the LOD.
  Challenge Phase Day 1: number analyzed (Participants) | 36 | 30
  Challenge Phase Day 1 | 76.2 [NA to NA] — The 95% confidence interval was not estimable as all samples were below the LOD. | 76.2 [NA to NA] — The 95% confidence interval was not estimable as all samples were below the LOD.
  Challenge Phase Day 2: number analyzed (Participants) | 66 | 55
  Challenge Phase Day 2 | 255.1 [143.9 to 452.1] | 341.2 [165.6 to 702.7]
  Challenge Phase Day 3: number analyzed (Participants) | 68 | 49
  Challenge Phase Day 3 | 6238.9 [2230.9 to 17447.5] | 15833.5 [5555.2 to 45129.2]
  Challenge Phase Day 4: number analyzed (Participants) | 49 | 40
  Challenge Phase Day 4 | 1970.7 [637.9 to 6088.1] | 16834.9 [4817.1 to 58834.9]
  Challenge Period Day 5: number analyzed (Participants) | 25 | 18
  Challenge Period Day 5 | 5412.0 [1150.7 to 25454.6] | 31096.5 [4975.1 to 194366.0]
  Challenge Phase Day 6: number analyzed (Participants) | 2 | 2
  Challenge Phase Day 6 | 1268.7 [0.0 to 4.2004828*10^18] | 4483.0 [0.1 to 207897355.4]
  Challenge Phase Day 8: number analyzed (Participants) | 75 | 64
  Challenge Phase Day 8 | 627.3 [340.0 to 1157.1] | 2737.3 [1400.4 to 5350.3]

17. Secondary Outcome: Geometric Mean GCs of NoV Shedding in Emesis Measured by qRT-PCR
Description: NoV shedding was assessed by qRT-PCR. Emesis samples were reported in 10^3 copies/mL. If a participant produced multiple results for a given study day, the result with the largest shedding response was used for analysis. Samples that were reported as "Not Quantifiable" or as lower than the limit of detection (LOD) were analyzed as ½2*LOD (15.3).
Time Frame: Pre-challenge up to Day 8 of Challenge Phase (equal to Study Day 36)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: 10^3 copies/mL
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 25 | 26
10^3 copies/mL
  Pre-challenge: number analyzed (Participants) | 0 | 0
  Challenge Phase Day 1: number analyzed (Participants) | 0 | 0
  Challenge Phase Day 2: number analyzed (Participants) | 12 | 15
  Challenge Phase Day 2 | 58.4 [19.8 to 172.4] | 457.3 [110.2 to 1897.5]
  Challenge Phase Day 3: number analyzed (Participants) | 20 | 26
  Challenge Phase Day 3 | 74.5 [24.9 to 222.7] | 152.5 [43.9 to 530.3]
  Challenge Phase Day 4: number analyzed (Participants) | 1 | 1
  Challenge Phase Day 4 | 15.3 [NA to NA] — The 95% confidence interval was not estimable as all samples were below the LOD and as only 1 participant was included. | 15.3 [NA to NA] — The 95% confidence interval was not estimable as all samples were below the LOD and as only 1 participant was included.
  Challenge Phase Day 5: number analyzed (Participants) | 2 | 1
  Challenge Phase Day 5 | 15.3 [NA to NA] — The 95% confidence interval was not estimable as all samples were below the LOD. | 15.3 [NA to NA] — The 95% confidence interval was not estimable as all samples were below the LOD and as only 1 participant was included.
  Challenge Phase Day 6: number analyzed (Participants) | 0 | 0
  Challenge Phase Day 8: number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Duration of NoV Infection
Description: Duration of NoV Infection was defined as the time from NoV infection to the time of resolution of infection, defined as a negative qRT-PCR result not followed by a positive qRT-PCR result.
Time Frame: Up to approximately Day 57
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 76 | 65
Hours | 120.1 [113.4 to 126.4] | 115.8 [109.5 to 122.2]

19. Other Pre Specified Outcome: VP1 GI.1-specific Fecal IgA at Day 1, Day 28 and Day 57
Description: Fecal samples for immunogenicity assessments were collected on Day 1 (prior to vaccination), Day 28 (1 day prior to challenge), and Day 57 (28 days post-challenge). VP1 GI.1-specific IgA antibody values were normalized by the total IgA in each sample.
Time Frame: Day 1 (baseline), Day 28 and Day 57
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mg
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 76 | 65
μg/mg
  Day 1 | 715.61 [442.64 to 1156.92] | 470.86 [316.78 to 699.89]
  Day 28 | 1888.49 [1221.06 to 2920.74] | 444.31 [304.83 to 647.60]
  Day 57: number analyzed (Participants) | 75 | 63
  Day 57 | 6122.41 [3891.96 to 9631.10] | 5047.07 [3000.20 to 8490.39]

20. Other Pre Specified Outcome: VP1 GI.1-specific Saliva IgA at Day 1, Day 28 and Day 57
Description: Saliva samples were collected on Day 1 (prior to vaccination), Day 28 (1 day prior to challenge), and Day 57 (28 days post-challenge). VP1 GI.1-specific IgA antibody values were normalized by the total IgA in each sample.
Time Frame: Day 1 (baseline), Day 28 and Day 57
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mg
Arm/Group | VXA-G1.1-NN | Placebo
Number analyzed (Participants) | 76 | 65
μg/mg
  Day 1 | 0.40 [0.31 to 0.51] | 0.31 [0.27 to 0.35]
  Day 28 | 1.15 [0.84 to 1.57] | 0.35 [0.31 to 0.40]
  Day 57: number analyzed (Participants) | 76 | 64
  Day 57 | 1.81 [1.33 to 2.44] | 1.84 [1.41 to 2.40]

ADVERSE EVENTS:
Time Frame: Up to approximately 16 months
Description: Safety Population: consisted of all participants who received any study vaccination (active or placebo). This population was summarized according to the actual vaccination received.
Arm/Group | VXA-G1.1-NN | Placebo
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/86 | 1/79
Other Adverse Events (participants affected / at risk) | 55/86 | 47/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VXA-G1.1-NN (N=86) | Placebo (N=79)
Deep vein thrombosis (Vascular disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VXA-G1.1-NN (N=86) | Placebo (N=79)
Abdominal pain (Gastrointestinal disorders) | 14 | 8
Diarrhoea (Gastrointestinal disorders) | 20 | 12
Nausea (Gastrointestinal disorders) | 13 | 10
Malaise (General disorders) | 25 | 20
Decreased appetite (Metabolism and nutrition disorders) | 10 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 12
Headache (Nervous system disorders) | 34 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT05212168/Prot_SAP_000.pdf